CLINICAL TRIAL: NCT06380959
Title: The Effects of Art-based Activities on Hope and Self-efficacy in Stroke Patients
Brief Title: Art-based Activities in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Esra Oksel, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 223K879
Record Dates: First submitted 2024-04-06; First posted 2024-04-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Stroke
Keywords: stroke; art therapy; Self-efficacy; Hope
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomised Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Based Activity Group (Experimental): The art-based activity module consists of 3 activities planned for 7 days.
  Interventions: Other: Art Based Activity
- Control Group (No Intervention): No intervention

INTERVENTIONS:
Other: Art Based Activity — Art Based Activity Module consists of 3 art-based activities under the titles "My Life Journey", "The Power Within Me" and "Letter to the Future". Each activity consists of three stages. In the first stage, the participants were made to practice breathing exercises. At this stage, the participant was expected to become aware of himself and his ideas. In the second stage, art activity was carried out. In the final stage, the revealed art object was concretized by the participants with a verbal expression. The materials used in the activities (dry paint, pastel paint, watercolor) are dermatologically tested and consist of anti-allergen products.
  Arms: Art Based Activity Group

SUMMARY:
Introduction and Aim: Life after stroke begins a difficult period in which functional capacity is very limited. Disability persists for a long time, and various problems such as hemiparesis, hemiplegia, dysarthria, dysphagia, urinary and bowel incontinence, which are frequently encountered after stroke, can affect the quality of life in the long term. As non-pharmacological approaches, especially non-invasive methods, have gained attention, creative arts-based therapies have often been recommended for stroke survivors because they have an arts-based approach without side effects. It is thought that the study conducted will contribute to the literature as there are not many studies in the literature. The aim of this study is to examine the effects of art-based activities on stroke patients' hope and self-efficacy levels. Its sub-purpose is to reveal the feelings and thoughts that arise with art objects obtained from art-based activities applied to stroke patients.

Materials and Methods: The study was conducted as a randomised controlled design. After the groups were determined, art-based activities module was applied to the intervention group for one week, while no additional intervention was made to the control group. Research data were collected using "Individual Introduction Form", "Herth Hope Index", "Generalized Self-Efficacy Scale. Data were analyzed with Statistical Package for the Social Sciences 25.0 package program. Written permission was obtained from the relevant ethics committee, hospital and participants to conduct the study.

DETAILED DESCRIPTION:
Introduction and Aim: Life after stroke begins a difficult period in which functional capacity is very limited. Disability persists for a long time, and various problems such as hemiparesis, hemiplegia, dysarthria, dysphagia, urinary and bowel incontinence, which are frequently encountered after stroke, can affect the quality of life in the long term. As non-pharmacological approaches, especially non-invasive methods, have gained attention, creative arts-based therapies have often been recommended for stroke survivors because they have an arts-based approach without side effects. It is thought that the study conducted will contribute to the literature as there are not many studies in the literature. The aim of this study is to examine the effects of art-based activities on stroke patients' hope and self-efficacy levels. Its sub-purpose is to reveal the feelings and thoughts that arise with art objects obtained from art-based activities applied to stroke patients.

Materials and Methods: The study was conducted as a randomised controlled design. After the groups were determined, art-based activities module was applied to the intervention group for one week, while no additional intervention was made to the control group. This research was conducted at the Neurology Clinic of Health Sciences University Izmir Bozyaka Training and Research Hospital between October 2023 and February 2024. The participants consisted of 72 patient 36 in the invention group and 36 in the control group with Modified Rankin Scale scores of 2 and 3 who were hospitalized with a stroke diagnosis in the Neurology Clinic. Research data were collected using "Individual Introduction Form", "Herth Hope Index", "Generalized Self-Efficacy Scale. Data were analyzed with Statistical Package for the Social Sciences 25.0 package program. Written permission was obtained from the relevant ethics committee, hospital and participants to conduct the study.

This study was supported by Scientific and Technological Research Council of Turkey (TUBITAK) under the Grant Number 223K879.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with a stroke
* Having a Modified Rankin Scale score of 2 and 3
* Not having plegia in the dominant hemisphere
* Not having a communication problem (cognitive, affective and verbal problems, etc.)
* Not having any disease that affects decision-making processes (dementia and psychiatric disease, etc.)
* Agreeing to participate in research

Exclusion Criteria:

• Refusing to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Herth Hope Index | Day 1 and Day 7
  It is a scale developed to measure the level of hope. The index consists of a 12-item Likert-type scale. This 4-point likert-type scale index assesses adults' general level of hope. Each item is scored on a scale from 1 (strongly disagree) to 4 (strongly agree), with a total score ranging from 12 to 48. The higher the score, the higher the level of hope.
Generalized Self-Efficacy Scale | Day 1 and Day 7
  It is a scale developed to measure the level of self-efficacy. The scores that can be obtained from the scale range from 10 to 40. An increase in the score indicates a higher level of self-efficacy in the individual.
Individual Introduction Form | Baseline
  This form was prepared by the researcher and includes questions regarding the sociodemographic and disease characteristics of the patients.

SECONDARY OUTCOMES:
Art Object Concretization Form | Day 2, Day 4 and Day 6
  It was created to concretize the unearthed art object through verbal expression. It contains a single open-ended question. After the art-based activity, the question was asked what the resulting art object meant.

CONTACTS AND LOCATIONS:
Overall Officials: Esra OKSEL, PhD, Study Director — Ege University
Locations (1):
- Ege University, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629